CLINICAL TRIAL: NCT05376293
Title: Web-based Intervention for Increasing Physical Activity in Cancer Survivors
Brief Title: Be-Active Study - Increasing Physical Activity in Cancer Survivors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Miriam Hospital (Other)
Collaborators: Brown University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1850077
Record Dates: First submitted 2022-05-06; First posted 2022-05-17 (Actual); Results first posted 2025-04-24 (Actual); Last update posted 2025-04-24 (Actual); Status verified 2025-01

CONDITIONS: Physical Activity; Exercise; Cancer Survivors
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Behavioral internet program (Active Comparator): Participants randomized to the Internet program will receive a 12-week behavioral Internet program designed to increase physical activity to recommended levels.
  Interventions: Behavioral: Behavioral Internet program
- Informational newsletter condition (Sham Comparator): Participants randomized to the newsletter condition will receive 6 newsletters, delivered every other week during the 3-month program.
  Interventions: Behavioral: Informational newsletter condition

INTERVENTIONS:
Behavioral: Behavioral Internet program — The 12-week behavioral Internet program is designed to increase physical activity to recommended levels. Participants will be asked to plan and report aerobic exercise weekly, watch weekly video lessons, and complete brief weekly homework assignments.
  Arms: Behavioral internet program
Behavioral: Informational newsletter condition — Newsletters will focus on the health benefits of regular physical activity, exercise safety, and will provide information on national exercise guidelines.
  Arms: Informational newsletter condition

SUMMARY:
Rates of cancer survivorship are on the rise and cancer survivors face unique health challenges that are common across cancer types that last well beyond the cessation of cancer treatment (e.g., increased fatigue, anxiety/depression, fear of recurrence, risk of cardiovascular disease, and lower health-related quality of life). While physical activity (PA) has favorable effects on these health parameters and is highly recommended for cancer survivors, this population engages in lower-than-average levels of PA. Effective PA interventions with high translation potential are important for improving the health of this population. The Internet overcome barriers to traditional face-to-face treatment programs (e.g., high cost, participant burden, geographical constraints) and represents a disseminable intervention approach. While behaviorally-based Internet programs significantly increase PA in other health domains, the application of these programs to cancer survivors is relatively new. This study will randomize 50 cancer survivors to a 12-week Internet PA program or usual-care newsletter condition. Primary outcomes include intervention engagement and program satisfaction related to the Internet program and changes in PA by intervention arm at post-treatment (3 months). Secondary aims include comparison of intervention arms on changes in sleep, weight, fatigue, anxiety/depression, health-related quality of life, and fear of recurrence.

ELIGIBILITY:
Inclusion Criteria:

* Confirmed cancer diagnosis and have either completed all cancer-directed treatment in the past 3-12 months or be on a maintenance/continuous treatment regimen for which they have been stable for at least 3 months
* Inactive - defined as engaging in <60 min/week of moderate-intensity PA over the past 3 months
* BMI between 18.5 and 45 kg/m2
* English speaking
* Daily Internet access

Exclusion Criteria:

* Any medical condition for which physical activity is contraindicated
* Unable to attend assessment visits in Providence RI

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-08-23 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2024-04-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- The Miriam Hospital's Weight Control and Diabetes Research Center, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- Behavioral Internet Program: Participants randomized to the Internet program received a 12-week behavioral Internet program designed to increase physical activity to recommended levels.
  Behavioral Internet program: The 12-week behavioral Internet program is designed to increase physical activity to recommended levels. Participants are asked to plan and report aerobic exercise weekly, watch weekly video lessons, and complete brief weekly homework assignments.
- Informational Newsletter Condition: Participants randomized to the newsletter condition receive 6 newsletters, delivered every other week during the 3-month program.
  Informational newsletter condition: Newsletters focus on the health benefits of regular physical activity, exercise safety, and provide information on national exercise guidelines.
Period: Overall Study
Arm/Group | Behavioral Internet Program | Informational Newsletter Condition
Started | 23 | 23
Completed | 22 | 22
Not Completed | 1 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Behavioral Internet Program | Informational Newsletter Condition | Total
Number analyzed (Participants) | 23 | 23 | 46
Age, Continuous [Mean (Standard Deviation); unit: years] | 54.4 (7.9) | 56.0 (8.8) | 55.2 (8.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 42
  Male | 4 | 0 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 4 | 5
  Not Hispanic or Latino | 22 | 19 | 41
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 1 | 2 | 3
  White | 20 | 18 | 38
  More than one race | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0

OUTCOME MEASURES:

1. Primary Outcome: Change in Physical Activity
Description: Change in minutes/week of moderate-to-vigorous intensity physical activity from baseline to 3 months as assessed by Actigraph accelerometers. Positive number indicates an increase in physical activity
Time Frame: baseline to 3 months
Measure: Mean (Standard Deviation); unit: minutes per week
Arm/Group | Behavioral Internet Program | Informational Newsletter Condition
Number analyzed (Participants) | 22 | 22
minutes per week | 49.3 (90.5) | 15.1 (100.4)

2. Primary Outcome: Intervention Engagement - Planning of Physical Activity (Internet Program Only)
Description: Participants were asked to submit an exercise plan (i.e., when they intended to exercise that week) at the beginning of weeks 2-12. This is the percentage of weeks that an exercise plan was submitted on the study website by the participant.
Time Frame: weekly from weeks 2-12
Measure: Mean (Standard Deviation); unit: percentage of weeks
Arm/Group | Behavioral Internet Program
Number analyzed (Participants) | 23
percentage of weeks | 82.6 (25.8)

3. Primary Outcome: Intervention Engagement - Self-monitoring of Physical Activity (Internet Program Only)
Description: Participants were asked to log their exercise minutes each week on the study website. This is the percentage of weeks that exercise minutes were reported on the study website by the participant over the 12-week period.
Time Frame: weekly during weeks 1-12
Measure: Mean (Standard Deviation); unit: percentage of weeks
Arm/Group | Behavioral Internet Program
Number analyzed (Participants) | 23
percentage of weeks | 85.9 (22.1)

4. Primary Outcome: Program Satisfaction Via Likert Scale
Description: Participants used a 1-7 Likert scale to answer 'how satisfied are you with the program received?" (higher score indicates greater satisfaction)
Time Frame: 3 months
Population: Note: one participant who was randomized to the Internet program only completed the primary outcome measure (physical activity), resulting in a sample of n=21 instead of n=22 for this measure.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Internet Program | Informational Newsletter Condition
Number analyzed (Participants) | 21 | 22
units on a scale | 5.81 (1.6) | 3.23 (1.6)

5. Secondary Outcome: Fatigue Measured Via the Brief Fatigue Inventory (BFI)
Description: The Brief Fatigue Inventory (BFI) assesses the severity of fatigue and the impact of fatigue on daily functioning. An overall fatigue score was calculated as the average of all answered items (range: 0-10) , with higher scores indicating more severe fatigue. Change in BFI score from baseline to 3 months was then calculated (a negative change scores indicates a reduction in fatigue).
Time Frame: baseline to 3 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Internet Program | Informational Newsletter Condition
Number analyzed (Participants) | 21 | 22
units on a scale | -0.32 (1.93) | -0.38 (1.91)

6. Secondary Outcome: Health-related Quality of Life (General Health Subscale) Measured Via the SF-36
Description: The 'General Health' subscale of the Short Form Health Survey (SF-36) evaluates a person's overall perception of their health. Scores range from 0 to 100, with higher scores indicating better perceived general health. Change scores from baseline to 3 months were then calculated (positive change scores indicate improved general health).
Time Frame: baseline to 3 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Internet Program | Informational Newsletter Condition
Number analyzed (Participants) | 21 | 22
units on a scale | 2.05 (10.54) | 3.64 (11.57)

7. Secondary Outcome: Psychological Distress Measured Via the 'Global Severity Index' Scale of the Brief Symptom Inventory-18 (BSI-18)
Description: Psychological distress was assessed using the 'Global Severity Index' of the Brief Symptom Inventory-18 (BFI-18). Scores range from 0 to 72, with greater scores indicating greater psychological distress. Change in psychological distress from baseline to 3 months was then calculated, with positive change scores indicating increased severity of symptoms such as somatization, depression, and anxiety.
Time Frame: baseline to 3 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Internet Program | Informational Newsletter Condition
Number analyzed (Participants) | 21 | 22
units on a scale | 0.1 (9.71) | 0.5 (5.18)

8. Secondary Outcome: Fear of Recurrence Measured Via the Fear of Cancer Recurrence Inventory (FCRI)
Description: A total score from the Fear of Recurrence Inventory - Short Form was used to assess the intensity of fear related to the possibility of cancer returning. Scores range from 0 to 36, with higher scores reflecting a greater severity of fear of cancer recurrence. Change scores from baseline to 3 months were then calculated (negative change scores indicates reduced fear of cancer recurrence)
Time Frame: baseline to 3 months
Population: as for outcome 4
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Behavioral Internet Program | Informational Newsletter Condition
Number analyzed (Participants) | 21 | 22
units on a scale | -1.67 (4.55) | -1.41 (4.33)

ADVERSE EVENTS:
Time Frame: Data were collected over the 3-month intervention period.
Description: Participants were instructed to inform the research staff if they had any injury or illnesses throughout the intervention period. Further, at the 3-month assessment visit, participants were queried regarding any potential adverse events over the past 3 months.
Arm/Group | Behavioral Internet Program | Informational Newsletter Condition
All-Cause Mortality (participants affected / at risk) | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/23 | 0/23
Other Adverse Events (participants affected / at risk) | 0/23 | 0/23

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-10-28): https://cdn.clinicaltrials.gov/large-docs/93/NCT05376293/Prot_000.pdf
  • Statistical Analysis Plan (2024-10-01): https://cdn.clinicaltrials.gov/large-docs/93/NCT05376293/SAP_001.pdf